CLINICAL TRIAL: NCT02037477
Title: Phase 3 Open-Label Crossover Pharmacodynamic Study to Evaluate the Acid-inhibitory Effect of TAK-438 20 mg With Esomeprazole 20 mg or Rabeprazole Sodium 10 mg in Healthy Adult Male Subjects
Brief Title: Phase 3 Study to Evaluate the Acid-Inhibitory Effect of Multiple Oral Doses of Vonoprazan (TAK-438)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAK-438/CPH-010; U1111-1152-3926 (Registry Identifier: UTN (WHO)); NCT02037477 (Registry Identifier: Clinicaltrials.gov); JapicCTI-142411 (Registry Identifier: JapicCTI); JapicCTI-R150821 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Esomeprazole; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence A (Cohort 1): Vonoprazan + Esomeprazole (Experimental): Vonoprazan (TAK-438) 20 mg, orally, once daily for 7 days, followed by a washout period of at least 7 days; then esomeprazole 20 mg, orally, once daily for 7 days.
  Interventions: Drug: Vonoprazan; Drug: Esomeprazole
- Sequence B (Cohort 1): Esomeprazole + Vonoprazan (Experimental): Esomeprazole 20 mg, orally, once daily for 7 days, followed by a washout period of at least 7 days; then vonoprazan 20 mg, orally, once daily for 7 days.
  Interventions: Drug: Vonoprazan; Drug: Esomeprazole
- Sequence C (Cohort 2): Vonoprazan + Rabeprazole Sodium (Experimental): Vonoprazan 20 mg, orally, once daily for 7 days, followed by a washout period of at least 7 days; then Rabeprazole sodium 10 mg, orally, once daily for 7 days.
  Interventions: Drug: Vonoprazan; Drug: Rabeprazole sodium
- Sequence D (Cohort 2): Rabeprazole Sodium + Vonoprazan (Experimental): Rabeprazole sodium 10 mg, orally, once daily for 7 days, followed by a washout period of at least 7 days; then vonoprazan 20 mg, orally, once daily for 7 days.
  Interventions: Drug: Vonoprazan; Drug: Rabeprazole sodium

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan tablets
  Other Names: TAK-438; Takecab®
Drug: Esomeprazole — Esomeprazole capsules
  Other Names: Nexium (esomeprazole)
  Arms: Sequence A (Cohort 1): Vonoprazan + Esomeprazole; Sequence B (Cohort 1): Esomeprazole + Vonoprazan
Drug: Rabeprazole sodium — Rabeprazole sodium tablets
  Other Names: Pariet (rabeprazole)
  Arms: Sequence C (Cohort 2): Vonoprazan + Rabeprazole Sodium; Sequence D (Cohort 2): Rabeprazole Sodium + Vonoprazan

SUMMARY:
The purpose of this study is to investigate the acid-inhibitory effect of multiple oral doses of Vonoprazan (TAK-438) and the relative effect of vonoprazan versus two controls (esomeprazole and rabeprazole sodium) in healthy Japanese adult male participants with the CYP2C19 extensive metabolizer (EM) genotype.

DETAILED DESCRIPTION:
This is a Phase 3 open-label crossover study to evaluate the acid-inhibitory effect following 7 days multiple doses of vonoprazan (20 mg per dose) and esomeprazole (20 mg per dose) (Cohort 1) or vonoprazan (20 mg per dose) and rabeprazole sodium (10 mg per dose) (Cohort 2) in healthy Japanese adult male participants (CYP2C19 genotype: EM). There will be a total of 20 participants, 5 per group for both Cohorts 1 and 2. At least 2 participants each with the homo EM (*1/*1) or hetero EM (*1/*2, *1/*3) CYP2C19 genotype will be enrolled among the 5 participants per group.

The drug being tested in this study is called vonoprazan. This study will look at the acid inhibitory effect following 7 days multiple doses of vonoprazan and esomeprazole (Cohort 1) or vonoprazan and rabeprazole sodium (Cohort 2) in healthy Japanese adult male participants with the CYP2C19 EM genotype.

The study will enroll a total of 20 participants, 5 per group for both Cohorts. At least 2 participants each with the homo EM (*1/*1) or hetero EM (*1/*2, *1/*3) CYP2C19 genotype will be enrolled among the 5 participants per group.

* Group A, Cohort 1: vonoprazan (20 mg per dose for 7 days) followed by esomeprazole (20 mg per dose for 7 days)
* Group B, Cohort 1: esomeprazole (20 mg per dose for 7 days) followed by TAK-438 (20 mg per dose for 7 days)
* Group C, Cohort 2: vonoprazan (20 mg per dose for 7 days) followed by rabeprazole sodium (10 mg per dose for 7 days)
* Group D, Cohort 2: rabeprazole sodium (10 mg per dose for 7 days) followed by vonoprazan (20 mg per dose for 7 days).

All participants will be asked to take Study Medication at the same time each day throughout the study. This single center trial will be conducted in Japan. The overall time to participate in this study is 31 days.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy Japanese adult male volunteer.
2. Is aged 20 to 45 years, inclusive, at the time of informed consent.
3. Has been confirmed at CYP2C19 genotyping as an Extensive Metabolizer [EM (*1/*1,*1/*2,*1/*3)].
4. Capable of understanding and complying with the protocol requirements.
5. The participant signs and dates a written informed consent form prior to the initiation of any study procedures.
6. Weighs 50 kg or more and has body mass index (BMI) of 18.5 or more and less than 25.0 kg/m^2 at Screening or admission (Day -3).
7. H. pylori-negative at Screening.

Exclusion Criteria:

1. Has undergone resection of the upper gastrointestinal tract or vagotomy.
2. Was determined to have hypoacidity or anacidity.
3. Has a present or past history of acid-related disease (reflux esophagitis, gastric ulcer, duodenal ulcer, non-erosive gastroesophageal reflux, Barrett's esophagus, Zollinger-Ellison syndrome, etc.).
4. Has undergone eradication of H. pylori within 6 months prior to the start of the study drug administration.
5. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormalities which may impact the ability of the subject to participate or potentially confound the study results.
6. Has a known hypersensitivities or allergies to drugs or food.
7. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 5 years prior to the start of the study drug administration.
8. Has poor peripheral venous access.
9. Had 200 mL or more of whole blood drawn within 4 weeks (28 days) prior to the start of the study drug administration or 400 mL or more of whole blood drawn within 12 weeks (84 days) prior to the start of the study drug administration.
10. Had a total volume of 800 mL or more of whole blood drawn within 52 weeks (364 days) prior to the start of the study drug administration.
11. Has undergone blood component draw within 2 weeks (14 days) prior to the start of the study drug administration.
12. Requires treatment with any of the excluded medications specified in the study or requires nutrition with any vitamin supplements or foods prohibited in the study.
13. Has received study medication within 16 weeks (112 days) prior to the start of the study drug administration.
14. Has received vonoprazan (TAK-438) in the past.
15. Has a history of cancer.
16. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen or serological reaction for syphilis at Screening.
17. Has a Screening or admission (Day -3) abnormal clinically significant electrocardiogram (ECG).
18. Has abnormal Screening or admission (Day -3) laboratory values that suggest a clinically significant underlying disease or subject with the following lab abnormalities: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > twice the upper limit of the normal range.
19. Is an immediate family member, study site employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
20. Participant who, in the opinion of the investigator or sub-investigator, is unlikely to comply with the protocol or is unsuitable for any other reasons.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Takeda
Locations (1):
- Fukuoka, Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 3 February 2014 to 27 March 2014.
Pre-assignment Details: A total of 56 participants signed the informed consent form. 20 participants were enrolled and received the study drug. The primary reason for ineligibility to receive the study drug was "did not meet entrance criteria" for 16 subjects. Nineteen subjects completed the study, while 1 subject withdrew due to a "pretreatment event/AE."
Groups:
- Sequence A (Cohort 1): Vonoprazan + Esomeprazole: Vonoprazan (TAK-438) 20 mg, orally, once daily for 7 days, followed by a washout period of at least 7 days and then esomeprazole 20 mg, orally, once daily for 7 days.
- Sequence B (Cohort 1): Esomeprazole + Vonoprazan: Esomeprazole 20 mg, orally, once daily for 7 days, followed by a washout period of at least 7 days and then vonoprazan 20 mg, orally, once daily for 7 days.
- Sequence C (Cohort 2): Vonoprazan + Rabeprazole Sodium: Vonoprazan 20 mg, orally, once daily for 7 days, followed by a washout period of at least 7 days and then rabeprazole sodium 10 mg, orally, once daily for 7 days.
- Sequence D (Cohort 2): Rabeprazole Sodium + Vonoprazan: Rabeprazole sodium 10 mg, orally, once daily for 7 days, followed by a washout period of at least 7 days and then vonoprazan 20 mg, orally, once daily for 7 days.
Period: Treatment Period 1
Arm/Group | Sequence A (Cohort 1): Vonoprazan + Esomeprazole | Sequence B (Cohort 1): Esomeprazole + Vonoprazan | Sequence C (Cohort 2): Vonoprazan + Rabeprazole Sodium | Sequence D (Cohort 2): Rabeprazole Sodium + Vonoprazan
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 1 | 0
Not completed — Pre-treatment Event/Adverse Event | 0 | 0 | 1 | 0
Period: Treatment Period 2
Arm/Group | Sequence A (Cohort 1): Vonoprazan + Esomeprazole | Sequence B (Cohort 1): Esomeprazole + Vonoprazan | Sequence C (Cohort 2): Vonoprazan + Rabeprazole Sodium | Sequence D (Cohort 2): Rabeprazole Sodium + Vonoprazan
Started | 5 | 5 | 4 | 5
Completed | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A (Cohort 1): Vonoprazan + Esomeprazole | Sequence B (Cohort 1): Esomeprazole + Vonoprazan | Sequence C (Cohort 2): Vonoprazan + Rabeprazole Sodium | Sequence D (Cohort 2): Rabeprazole Sodium + Vonoprazan | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (6.93) | 23.8 (5.17) | 22.2 (2.95) | 25.2 (2.95) | 25.2 (5.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 5 | 5 | 5 | 5 | 20
Region of Enrollment [Number; unit: participants]
  Japan | 5 | 5 | 5 | 5 | 20
Height [Mean (Standard Deviation); unit: cm] | 172.0 (7.75) | 173.0 (6.52) | 172.8 (6.76) | 169.4 (4.88) | 171.8 (6.48)
Weight [Mean (Standard Deviation); unit: kg] | 64.10 (8.930) | 64.10 (9.813) | 62.68 (5.008) | 58.34 (5.227) | 62.31 (7.245)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.56 (1.674) | 21.32 (1.844) | 20.96 (0.808) | 20.34 (1.222) | 21.05 (1.387)
CPY2C19 Genotype Test (N) [Number; unit: participants]
  Homo Extensive Metabolizer (EM) | 2 | 3 | 3 | 2 | 10
  Hetero EM | 3 | 2 | 2 | 3 | 10
  Poor Metabolizer (PM) | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intragastric pH Time Course Over 24 Hours
Description: Intragastric pH was measured continuously for 24 hours (hr) by pH monitor. pH holding time ratio (HTR) is the percentage of time a pH is maintained at a particular level. For example, pH 4 HTR is the percentage of time the pH = 4.
Time Frame: At baseline (Day -2 to Day -1), administration period (Days 1 to Day 2 and Days 7 to Day 8)
Population: Pharmacodynamic (PD) Analysis Set - Participants receiving study medication who completed protocol procedures without serious violation of the protocol were eligible for PD analysis. All 10 subjects from Cohort 1 were included. Three subjects in Cohort 2 were excluded from the PD analysis set, which therefore consisted of 7 subjects.
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Cohort 1 - Vonoprazan 20 mg; Cohort 2 - Vonoprazan 20 mg: Vonoprazan 20 mg, orally, once daily for 7 days.
- Cohort 1 - Esomeprazole 20 mg: Esomeprazole 20 mg, orally, once daily for 7 days.
- Cohort 2 - Rabeprazole Sodium 10 mg: Rabeprazole sodium 10 mg, orally, once daily for 7 days.
Arm/Group | Cohort 1 - Vonoprazan 20 mg | Cohort 1 - Esomeprazole 20 mg | Cohort 2 - Vonoprazan 20 mg | Cohort 2 - Rabeprazole Sodium 10 mg
Number analyzed (Participants) | 10 | 10 | 7 | 7
percentage of time
  0-24 hr pH 4 HTR (%)-Baseline | 10.63 (7.391) | 10.63 (7.391) | 8.90 (6.472) | 8.90 (6.472)
  0-24 hr pH 4 HTR (%)-Day 1 | 71.37 (17.030) | 23.92 (16.896) | 84.16 (12.383) | 26.29 (13.381)
  0-24 hr pH 4 HTR (%)-Day 7 | 85.82 (14.748) | 61.21 (17.140) | 93.79 (7.310) | 65.09 (14.159)
  0-12 hr pH 4 HTR (%)-Baseline | 12.98 (11.139) | 12.98 (11.139) | 8.01 (5.730) | 8.01 (5.730)
  0-12 hr pH 4 HTR (%)-Day 1 | 74.83 (9.681) | 34.89 (24.645) | 84.03 (7.810) | 37.26 (20.384)
  0-12 hr pH 4 HTR (%)-Day 7 | 96.45 (4.402) | 77.62 (17.302) | 98.83 (2.968) | 76.06 (9.591)
  12-24 hr pH 4 HTR (%)-Baseline | 8.18 (13.735) | 8.18 (13.735) | 9.77 (14.096) | 9.77 (14.096)
  12-24 hr pH 4 HTR (%)-Day 1 | 67.86 (28.345) | 12.94 (10.876) | 84.34 (20.254) | 15.34 (13.317)
  12-24 hr pH 4 HTR (%)-Day 7 | 75.21 (26.398) | 44.81 (17.338) | 88.77 (14.369) | 54.13 (25.275)

2. Secondary Outcome: Frequency of Adverse Events
Description: The frequency of adverse events by type, seriousness, time to onset. Adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug to the last dose of study drug.
Time Frame: 31 days
Population: Safety analysis set - All participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1 - Vonoprazan 20 mg | Cohort 1 - Esomeprazole 20 mg | Cohort 2 - Vonoprazan 20 mg | Cohort 2 - Rabeprazole Sodium 10 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants
  Treatment Emergent Adverse Events | 0 | 0 | 3 | 1
  Related | 0 | 0 | 1 | 0
  Not Related | 0 | 0 | 2 | 1
  Mild | 0 | 0 | 2 | 1
  Moderate | 0 | 0 | 1 | 0
  Severe | 0 | 0 | 0 | 0
  Leading to Study Drug Discontinuation | 0 | 0 | 1 | 0

3. Secondary Outcome: Number of Participants With Abnormal Changes From Baseline in Vital Signs
Description: Vital signs included body temperature (oral or tympanic measurement), sitting blood pressure (after the participant has rested for at least 5 minutes), and pulse (bpm).
Time Frame: At screening, baseline (Day -3, Day -2, Day -1), administration period (Days 1, Day 2, Day 7, Day 8), and post-test (Day 28)
Population: Safety analysis set - All participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1 - Vonoprazan 20 mg | Cohort 1 - Esomeprazole 20 mg | Cohort 2 - Vonoprazan 20 mg | Cohort 2 - Rabeprazole Sodium 10 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (at Rest) Findings
Time Frame: At Screening, baseline (Day -3), administration period (Day 8), and post-test (Day 28)
Population: Safety analysis set - All participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1 - Vonoprazan 20 mg | Cohort 1 - Esomeprazole 20 mg | Cohort 2 - Vonoprazan 20 mg | Cohort 2 - Rabeprazole Sodium 10 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Markedly Abnormal Laboratory Values
Description: The number of participants with markedly abnormal laboratory values for Chemistry, Hematology and Urinalysis during the study is reported.
Time Frame: At Screening, baseline (Day -3), administration period (Day 1, Day 8), and post-test (Day 28)
Population: Safety analysis set - All participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1 - Vonoprazan 20 mg | Cohort 1 - Esomeprazole 20 mg | Cohort 2 - Vonoprazan 20 mg | Cohort 2 - Rabeprazole Sodium 10 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 31 Days
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1 - Vonoprazan 20 mg | Cohort 1 - Esomeprazole 20 mg | Cohort 2 - Vonoprazan 20 mg | Cohort 2 - Rabeprazole Sodium 10 mg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 3/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Vonoprazan 20 mg (N=10) | Cohort 1 - Esomeprazole 20 mg (N=10) | Cohort 2 - Vonoprazan 20 mg (N=10) | Cohort 2 - Rabeprazole Sodium 10 mg (N=10)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.